CLINICAL TRIAL: NCT01488253
Title: Multicenter Trials to Evaluate the Efficacy and Toxicity of Sirolimus/Tacrolimus Combination as a GVHD Prophylaxis After HLA Matched Related PBSCT
Brief Title: Sirolimus/Tacrolimus Combination After HLA Matched Related Peripheral Blood Stem Cell Transplants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We could not receive the support from the national medical insurance owing to the changed policy of the government for clincal trials.
Sponsor: The Korean Society of Blood and Marrow Transplantation (Other)
Collaborators: Asan Medical Center (Other); Chonbuk National University Hospital (Other); Chonnam National University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Daegu Catholic University Medical Center (Other); Ewha Womans University Mokdong Hospital (Other); Gachon University Gil Medical Center (Other); Inha University Hospital (Other); Inje University (Other); Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); Pusan National University Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); Seoul St. Mary's Hospital (Other); Seoul National University Hospital (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Seong Kyu Park, MD, Director of Clinical Trials Committee, The Korean Society of Blood and Marrow Transplantation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KSBMT2011-01
Record Dates: First submitted 2011-11-20; First posted 2011-12-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Acute Leukemia in Remission; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated-Phase
Keywords: Hematopoietic stem cell transplantation; Graft vs Host disease; Prevention; Sirolimus; Tacrolimus
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Graft vs Host Disease | interventions — Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- acute GVHD prevention by sirolimus based regimen (Experimental): The investigators will evaluated the primary endpoint and secondary endpoints comparing with historical control, that is used tacrolimus/methotrexate as a GVHD prophylaxis after HLA-matched, related PBSCT.
  Interventions: Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus will be administered as a 6-mg oral loading dose beginning on day -1, followed by 3 mg per day orally in a single morning dose with a target trough level of 5-12 ng/mL. Trough levels will be measured once a week. Sirolimus will be gradually tapered beginning at day +100, and eliminated by day +180, unless the patient required continued treatment for GVHD or experienced toxicity related to drugs.
  Other Names: Rapamune (sirolimus, rapamycin)
Drug: Tacrolimus — Tacrolimus will be administered beginning on day -1 at 0.05 mg/kg intravenously by continuous infusion every 24 hours, with a target serum level of 5 to 10 ng/mL. Tacrolimus dosing is converted to oral capsules prior to discharge. Trough levels will be measured once a week. Tacrolimus will be gradually tapered beginning at day +100, and eliminated by day +180, unless the patient required continued treatment for GVHD or experienced toxicity related to drugs.
  Other Names: Prograf (tacrolimus)

SUMMARY:
Study Design: To evaluate the efficacy of the combination of sirolimus and tacrolimus as a graft-versus-host disease prophylaxis, the investigators are going to perform a phase II, multicenter clinical trial after human leukocyte antigen (HLA)-matched, related peripheral blood stem cell transplants (PBSCT) in patients with hematologic malignancies. Total 116 patients will be accrued.

Objective: The primary objective is to evaluate the rates of 100 day Grade II-IV acute GVHD. Secondary objectives include the time to neutrophil and platelet engraftment, the incidence of grade III-IV acute GVHD, non-relapse mortality during 100 days after transplant, mucositis severity, all infectious complications including cytomegalovirus (CMV) reactivation, vascular complications (venoocclusive disease of liver; VOD, thrombotic microangiopathy; TMA), disease-free survival, and overall survival at 1 year after transplant.

Eligibility Criteria: Eligible patients are between 20 and 60 years of age, have acute leukemia, myelodysplastic syndrome (MDS), chronic myelogenous leukemia (CML), and adequate organ function. For available sibling donor, a serologic (or higher resolution) 6/6 Class I HLA-A and B and molecular Class II DRB1 must be matched.

Treatment Description: Conditioning regimens will vary by center and donor will donate peripheral blood stem cells according to local institutional practices. Peripheral blood stem cells will not be manipulated or T-depleted prior to infusion. Tacrolimus will be administered at 0.05 mg/kg/day intravenously by continuous infusion beginning on day -1 with a target serum concentration of 5 to 10 ng/mL. Sirolimus will be administered as a 6 mg oral loading dose on day -1, followed by a 3 mg/day single dose, with a target serum concentration of 3 to 12 ng/mL. Levels will be monitored weekly during hospitalization and then as clinically indicated. Intravenous tacrolimus will be converted to an oral equivalent dose prior to discharge and both immunosuppressives will be tapered beginning at day +100 after transplantation and eliminated by day +180 when clinically feasible.

Accrual Period: The estimated accrual period is three years. Patients will be followed for 100 days post transplantation for evaluation of the primary endpoint, with additional follow-up to two years after transplantation for evaluation of secondary endpoints.

DETAILED DESCRIPTION:
Rationale: Graft-versus-host disease (GVHD) remains a major cause of morbidity and mortality after allogeneic HSCT. The combination of a calcineurin inhibitor and methotrexate has been the standard GVHD prophylactic regimen for the past 20 years. However, the incidence of acute GVHD remains high, with reported cumulative incidence of grade II-IV up to 60%. Serious acute GVHD or chronic GVHD has detrimental consequences in patients including death, disability, infections, or prolonged hospitalization.

Sirolimus is the first available inhibitor of the mammalian target of rapamycin (mTOR). And sirolimus binds uniquely to FK-binding protein (FKBP12) and forms a complex with mTOR. This complex inhibits several biochemical pathways, resulting in a reduction in DNA transcription, DNA translation, protein synthesis, and cell cycling, ultimately leading to T-cell immunosuppression. Sirolimus has been used alone and in combination with calcineurin inhibitors for prevention of allograft rejection after solid organ transplantation. In the field of hematopoietic stem cell transplantation, the combination of sirolimus and tacrolimus has also resulted in a low incidence of acute GVHD and reduced transplant-related toxicity.

In addition, the investigators demonstrated previously that the combination of tacrolimus and sirolimus is effective as a GVHD prophylaxis and well tolerated in cases of high risk transplantation using mismatched related or unrelated donor.

As discussed above, sirolimus has emerged as one of the most promising immunosuppressive agents in allogeneic hematopoietic stem cell transplantation. However, the benefit of GVHD prophylaxis regimens including sirolimus has not been confirmed consistently and there is controversy that the incorporation of sirolimus into GVHD prophylaxis results in improved survival.

Efficacy measures: Patients will be followed for 100 days post transplantation for evaluation of the primary endpoint (the incidence and severity of acute GVHD) and clinical data will be collected at 100 day after HSCT using case report form. And patients will be recommended additional follow-up to one year after HSCT for evaluation of secondary endpoints or parameters including clinical outcomes (disease-free survival and overall at 1 year after transplant). The investigators will perform the interim analyses at the time when 31 patients are enrolled during phase 1.

Acute GVHD will be graded according to the consensus grading scale (appendix-1). The broad category of acute GVHD includes:

1. Classic acute GVHD (maculopapular rash, nausea, vomiting, anorexia, profuse diarrhea, illus, or cholestatic hepatitis) occurring within 100 days after transplantation (without diagnostic or distinctive signs of chronic GVHD)
2. Persistent, recurrent, or late acute GVHD: Features of classic acute GVHD without diagnostic or distinctive manifestations of chronic GVHD occurring beyond 100 days of transplantation (often seen after withdrawal of immune suppression).

Safety: All the safety analyses will be based on safety population. The assessment of safety will be based mainly on the frequency of adverse events and on the number of laboratory values that fall outside of predetermined ranges. Adverse events will be summarized by presenting the number and percentage of patients having any adverse event as well as by severity to study treatment. In addition the summary of grade 3 and 4 will be presented.

During administration of drugs as a GVHD prophylaxis, toxicities related to drugs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v3.0). Patients will also be assessed regularly by physical examination and laboratory tests including CBC, biochemistry including liver function test and chest X-ray.

Statistical Methods: Descriptive statistical analysis will be performed to assess patient baseline characteristics, engraftment, acute GVHD, and non-relapse mortality. Overall survival and relapse-free survival will be calculated using the Kaplan-Meier method and estimated using a competing risk of 100-day mortality for cumulative incidence rate of grades II-IV acute GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent prior to participating to the study
* Patients with acute leukemia in remission, MDS, and CML in chronic & accelerated phase
* Patients with HLA identical donor, a serologic (or higher resolution) 6/6 Class I HLA-A and B and molecular Class II DRB1 must be matched.
* Patients with an ECOG performance status score < 2
* Adequate end organ functions as defined by: Total bilirubin < 1.5 × ULN, AST and ALT < 2.5 × ULN, Creatinine < 1.5 × ULN.
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days before initiation of study drug.

Exclusion Criteria:

* Acute promyelocytic leukemia (M3)
* Patients with another primary malignancy other than hematologic disease
* Patients with a severe or uncontrolled medical condition (i.e. uncontrolled diabetes, chronic renal disease)
* Patients who are ① pregnancy, ② breast feeding, ③ of childbearing potential without a negative pregnancy test prior to baseline and ④ male or female of childbearing potential unwilling to use barrier contraceptive precautious throughout the trial (post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential)
* Patients with an ECOG performance status score ≥ 2
* Patients with known positivity for HIV; baseline testing for HIV is not required

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The rate of grade II-IV acute graft-versus host disease | 100 days after allogeneic HSCT
  Patients will be followed for 100 days post transplantation for evaluation of the primary endpoint (the incidence and severity of acute GVHD) and clinical data will be collected at 100 day after HSCT using case report form. Acute GVHD will be graded according to the consensus grading scale.

SECONDARY OUTCOMES:
The time to neutrophil and platelet engraftment | within 6 weeks after transplant
  The time of engraftment is defined as the first of three consecutive days on which the absolute neutrophil counts exceed 0.5 X 10(9)/L and platelet count to 20 X 10(9)/L, respectively.
The incidence of grade III-IV acute GVHD | During 100 days after transplant
  Acute GVHD will be graded according to the consensus grading scale.
Non-relapse mortality | During 100 days after transplant
  All deaths without relapse or progression of underlying disease
Mucositis severity | 100 days after transplant
  It will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v3.0).
All infectious complications including CMV reactivation | 100 days after transplant
  The incidence and type of infectious complications
Vascular complications | 100 days after transplant
  The incidence of venoocclusive disease of liver and syndrome of thrombotic microangiopathy.
Clinical outcome at 1 year after transplant | 1 year after transplant
  Disease-free survival and overall survival at 1 year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Seong Kyu Park, MD, PhD, Principal Investigator — Clinical Trials Committee of The Korean Society of Blood and Marrow Transplantation
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea